CLINICAL TRIAL: NCT04022135
Title: Is Natural Folate as Effective as Synthetic Folic Acid in Increasing Serum and Red Blood Cell Folate Concentrations During Pregnancy? A Proof-of-concept Pilot Study
Brief Title: Natural Folate vs. Synthetic Folic Acid in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: BC Children's Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Crystal Karakochuk, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: H18-02635
Record Dates: First submitted 2019-07-14; First posted 2019-07-16 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Pregnancy
Keywords: folate; folic acid; nutrition; pregnancy
MeSH Terms: interventions — Folic Acid; levomefolate calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Folic acid (Active Comparator): 0.6 mg/day
  Interventions: Dietary Supplement: Folic acid
- (6S)-5-methyltetrahydrofolic acid (Metafolin) (Experimental): 0.625 mg/d (an equimolar dose to folic acid)
  Interventions: Dietary Supplement: (6S)-5-methyltetrahydrofolic acid

INTERVENTIONS:
Dietary Supplement: Folic acid — Participants will supplement with 0.6mg/day for 16 weeks.
  Arms: Folic acid
Dietary Supplement: (6S)-5-methyltetrahydrofolic acid — Participants will supplement with 0.625mg/day for 16 weeks.
  Other Names: Metafolin
  Arms: (6S)-5-methyltetrahydrofolic acid (Metafolin)

SUMMARY:
In this two-arm, double-blind randomized pilot study, the investigators will recruit 60 generally healthy, low-risk pregnant women aged 19-42 years living in Vancouver, Canada. Participants will be randomized to supplement with either 0.6 mg/day folic acid or an equimolar dose (0.625 mg/day) of (6S)-5-methyltetrahydrofolic acid for 16-weeks of their pregnancy. Randomization will occur at 8-21 weeks gestation (after neural tube closure) to reduce the risk of harm should the natural folate prove less effective. All participants will also receive a prenatal multivitamin not containing any form of folate, to ensure adequacy of other nutrients (e.g. iron) required during pregnancy. Three-hour fasting venous blood samples will be collected at baseline and endline to measure serum and red blood cell folate, unmetabolized folic acid and other related biomarkers. Women will be given the option to continue supplementing until 1-week postpartum, and provide a small (3mL) breastmilk sample and blood sample in order to measure differences in folates in breastmilk and postpartum folate. These pilot data will be used to inform a definitive trial regarding the most effective form of folate supplementation for mothers and their babies.

DETAILED DESCRIPTION:
A sample size of 50 women (25 in each group) are required to reliably estimate the distributions of serum and red blood cell folate. Thus, to account for drop outs or loss to follow up, a total of 60 women (30 in each group) will be recruited.

Aim 1: To establish the mean ± standard deviation change in serum folate, red blood cell folate, and unmetabolized folic acid levels in each group following supplementation with (6S)-5-methyltetrahydrofolic acid or folic acid for 16-weeks of pregnancy.

Aim 2: To determine participation recruitment and retention rate, the most effective recruitment strategies for this population, and adherence to study protocol (to inform a definitive trial).

Exploratory Aims: To explore differences in proposed clinical effects associated with folic acid supplementatation (immunity, gene methylation) and differences in biomarkers that function closely with folate in one carbon metabolism (B-vitamins, choline and its metabolites [betaine, dimethylglycine]) and which support overall blood health (ferritin, inflammation). In the postpartum phase, we will quantify proportion of total breastmilk folate as folic acid in each group, evaluate correlation of maternal postpartum plasma unmetabolized folic acid and breastmilk folic acid, and to evaluate RBC folate concentrations following delivery in each group. Differences in breastmilk biomarkers associated with folate (choline, human milk oligosaccharides, and breastmilk microbiome) will be explored.

Women may undergo informed consent process anytime <21 weeks gestation. Once participants indicate that they are interested in participating in the trial, the participant will be given a study ID, and a baseline visit will be scheduled.

The baseline visit will occur between 8-21 weeks gestation, and will involve discontinuation of current folate/prenatal vitamin supplementation, review and signing the informed consent form (a scanned copy will be shared with the participant), randomization to a folate group, provision of study supplements, completion of a baseline questionnaire, completion of a food frequency questionnaire, measurement of weight and height, and a small blood draw (12ml).

Intervention: total time: 16 weeks. Participants will supplement daily with the folate and prenatal vitamin supplements. The research coordinator will call the participants half way through the intervention period to serve as a reminder and answer any questions, which will enhance protocol adherence.

The endline visit will occur between 24-37 weeks gestation, and will involve collecting any remaining supplements (for capsule counts), a weight measurement, and a small blood draw (12ml), and completion of a short endline questionnaire.

Optional continuation of study: After the endline visit, women who are planning to breastfeed will have the option to continue supplementing with the study supplements until approximately 1 week postpartum, at which time they will provide a small (3 mL) breastmilk sample and/or blood sample.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman (singleton pregnancy)
* Living in the Greater Vancouver area and willing to travel to the University of British Columbia for study visits
* <21 weeks gestation
* 19-42 years of age
* willing to participate

Exclusion Criteria:

* Have a pre-existing medical condition known to impact maternal folate status (malabsorptive of irritable bowel disease, active celiac disease, gastric bypass surgery, atrophic gastritis, epilepsy, advanced liver disease, kidney dialysis, type 1 or 2 diabetes mellitus, sickle cell trait/anemia)
* Lifestyle factors known to impact maternal folate status (smoking, alcohol overuse, non-prescription drug use/abuse)
* Are medium to high risk for development of an NTD-affected pregnancy (applies to women or their male partner: personal or family history [parents or siblings] of other folate sensitive congenital anomalies, personal NTD history or a previous NTD-affected pregnancy)
* Are taking medications known to interfere with B-vitamin metabolism (Chloramphenicol, Methotrexate, Metformin, Sulfasalazine, Phenobarbital, Phenytoin, Primidone, Triamterene, Barbiturates)
* pre-pregnancy body mass index ≥30 kg/m2
* allergic to any of the supplement ingredients

Ages: 19 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-09-08 (Actual)

PRIMARY OUTCOMES:
Concentration of red blood cell folate levels | concentrations at both baseline (8-21 weeks gestation), endline (24-37 weeks gestation), and postpartum
  nmol/L; Reflects longer term status (e.g. previous 3-4 months)
Concentration of serum folate levels | concentrations at both baseline (8-21 weeks gestation), endline (24-37 weeks gestation), and postpartum
  nmol/L; Reflects recent status or dietary intake
Concentration of unmetabolized folic acid (and other folate forms: THF, 5-Methyl-THF, 5-formyl-THF, and 5,10-methenyl-THF) | concentrations at both baseline (8-21 weeks gestation), endline (24-37 weeks gestation), and postpartum
  nmol/L; unmetabolized folic acid is not incorporated into RBCs, rather it circulates in plasma

SECONDARY OUTCOMES:
Concentration of total vitamin B-12 | concentrations at both baseline (8-21 weeks gestation), endline (24-37 weeks gestation)
  pmol/mL; closely involved in folate metabolism and facilitating methionine cycles
Concentration of pyridoxal-5'-phosphate | concentrations at both baseline (8-21 weeks gestation), endline (24-37 weeks gestation)
  nmol/L; closely involved in folate metabolism and facilitating methionine cycles
Concentration of vitamin B2 | concentrations at both baseline (8-21 weeks gestation), endline (24-37 weeks gestation)
  nmol/L; closely involved in folate metabolism and facilitating methionine cycles
Concentration of betaine | concentrations at both baseline (8-21 weeks gestation), endline (24-37 weeks gestation)
  µmol/L; closely involved in facilitating methionine cycles
Concentration of choline | concentrations at both baseline (8-21 weeks gestation), endline (24-37 weeks gestation)
  µmol/L; closely involved in facilitating methionine cycles
Concentration of dimethylglycine | concentrations at both baseline (8-21 weeks gestation), endline (24-37 weeks gestation)
  µmol/L; closely involved in facilitating methionine cycles
Concentration of S-adenosyl-methionine | concentrations at both baseline (8-21 weeks gestation) and endline (24-37 weeks gestation)
  µM; Metabolite produced in methionine cycles
Concentration of S-adenosyl-homocysteine | concentrations at both baseline (8-21 weeks gestation) and endline (24-37 weeks gestation)
  µM; Metabolite produced in methionine cycles
Concentration of total homocysteine | concentrations at both baseline (8-21 weeks gestation) and endline (24-37 weeks gestation)
  µmol/L; Metabolite produced in methionine cycles
Concentration of methionine | concentrations at both baseline (8-21 weeks gestation) and endline (24-37 weeks gestation)
  µmol/L; Metabolite produced in methionine cycles
Concentration of cysteine | concentrations at both baseline (8-21 weeks gestation) and endline (24-37 weeks gestation)
  µmol/L; Metabolite produced in methionine cycles
Collection of peripheral blood mononuclear layer cells | Collection at both baseline (8-21 weeks gestation), endline (24-37 weeks gestation)
  Gene variant assessment of MTHFR (677 C>T, rs1801133, and 1298 A>C, rs1801131) and DHFR (rs1643649 and rs70991108) and differences in DNA methylation, and frequency and cytotoxicity of immune cells in PBMCs.
Concentration of unmetabolized folic acid in breastmilk (and other folate forms: THF, 5-Methyl-THF, 5-formyl-THF, and 5,10-methenyl-THF) | Collection at 1 week postpartum
  nmol/L; folic acid that is unmetabolized and enters breastmilk as such
Folate binding protein in breastmilk | Collection at 1 week postpartum
  nmol folate binding per liter of milk
Breastmilk fatty acids & choline forms (free choline, betaine, phosphocholine, glycerophosophocholine) | Collection at 1 week postpartum
  Quantified via LC-MS/MS
Breastmilk human milk oligosaccharides and breastmilk microbiome | Collection at 1 week postpartum
  Quantified via HPLC-FL and PCR
Complete blood count | Baseline (8-21 weeks gestation), endline (24-37 weeks gestation), and postpartum
  Analysis will be performed using an automated hematology analyzer (Sysmex XNL550, Kobe, Japan)
Markers of Iron and Inflammation | Baseline (8-21 weeks gestation),and endline (24-37 weeks gestation)
  This will include measurement of serum ferritin (µg/L), soluble transferrin receptor (mg/L), body iron stores (mg/kg), retinol binding protein (µmol/L), CRP (mg/L), and AGP (g/L) in serum using a sandwich ELISA, and hormones that influence iron regulation in pregnancy, including serum hecipdin (ng/mL; measured with an ELISA) and serum erythropoietin (mIU/mL; measured with an immunoassay)

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Karakochuk, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Food Nutrition and Health Building, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after de-identification, will be available immediately following publication. Anyone who is interested in accessing the data should send a proposal to the principal investigator for approval to gain access.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: All data will be available following publication for approximately 5 years after initial collection.
Access Criteria: A proposal from those interested in accessing the data should be sent to study investigators for access approval.

REFERENCES:
- [Derived] Cochrane KM, Hutcheon JA, Karakochuk CD. Iron-Deficiency Prevalence and Supplementation Practices Among Pregnant Women: A Secondary Data Analysis From a Clinical Trial in Vancouver, Canada. J Nutr. 2022 Oct 6;152(10):2238-2244. doi: 10.1093/jn/nxac135. PMID 35687377
- [Derived] Cochrane KM, Mayer C, Devlin AM, Elango R, Hutcheon JA, Karakochuk CD. Is natural (6S)-5-methyltetrahydrofolic acid as effective as synthetic folic acid in increasing serum and red blood cell folate concentrations during pregnancy? A proof-of-concept pilot study. Trials. 2020 May 5;21(1):380. doi: 10.1186/s13063-020-04320-3. PMID 32370802

DOCUMENTS (1):
  • Study Protocol (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/35/NCT04022135/Prot_001.pdf